CLINICAL TRIAL: NCT06105359
Title: The Effect of Dignity Therapy Applied to End-stage Cancer Patients on Perceived Dignity and Self-esteem: a Randomized Controlled Trial
Brief Title: The Effect of Dignity Therapy Applied to Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, NESIBE GÜNAY MOLU, Assoc. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Necmettin Erbakan University1
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Dignity
Keywords: Dignity therapy; cancer patient; depression
MeSH Terms: conditions — Neoplasms; Depression | interventions — Dignity Therapy

STUDY DESIGN:
Intervention Model Description: Research, experimental control group and pretest-posttest study will be carried out.
Who Masked: Participant, Outcomes Assessor
Masking Description: To control for performance bias, patients will be blinded to the study hypothesis and will not be informed which group they are in. There will be no blinding for the researcher. However, blind technique will be used in the research. This blind technique will be applied by the researcher with the patients blinded until the application begins. In the research, in order to meet the blind technical conditions, the process steps were carried out by an independent statistician from the first stage. The sample will be sorted by a combination order and number. In this way selection bias will be controlled. The study will also be controlled for attrition bias and Statistics and reporting bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients in this group will be treated with dignity therapy by the researcher.
  Interventions: Behavioral: Dignity therapy; Other: standardize care
- control group (Active Comparator): Patients in this group will receive standard care and no treatment will be performed by the researcher.
  Interventions: Other: standardize care

INTERVENTIONS:
Behavioral: Dignity therapy — Dignity therapy will be applied in the interview room that will be requested in the oncology clinic to protect the confidentiality of information.
  The application is planned as five sessions and the sessions will last approximately 40 minutes. Two questions in the dignity therapy protocol will be discussed in each session.
  Arms: experimental group
Other: standardize care — Patients in this group will receive standard treatment and care in the clinic. No action will be taken other than standard care.
  Other Names: Cancer patients will receive routine treatment and care.

SUMMARY:
The aim of this study is to determine the effect of dignity therapy on the quality of life and depression levels of cancer patients.

Methods: The research was planned as a randomized controlled experimental study.

Type of Research: Research, experimental, control group and pretest-posttest study will be carried out.

Population of the Study: The population of the study was sent to Meram Medical Faculty Hospital Oncology Clinic consists of male and female inpatients.

Sample of the Research: Those who agreed to participate in the research and met the inclusion criteria. Patients who meet will be included in the study. It was 48. It was planned to be.

Randomization: In this study, parallel group block randomization method was applied to the intervention and control groups. will be allocated randomly. Block randomization was used because the sample size was small. Patients will be selected equally using permutation method, and randomization will be selected using blocking technique. will be done. During randomization, CONSORT 2017 will be used.

For randomization; To control for performance bias, patients will be blinded to the study hypothesis and will not be informed which group they are in. There will be no blinding for the researcher. However, blind technique will be used in the research. This blind technique will be applied by the researcher with the patients blinded until the application begins..

Data Collection Techniques and Tools: "Personal Information Form", "Patient Dignity Inventory" and "Rosenberg Self-Esteem Scale" were used in data collection (RSES)" will be used.

DETAILED DESCRIPTION:
Cancer affects both the patient and their relatives physically and psychologically. From the moment cancer is diagnosed, psychological problems that affect the adaptation processes of individuals, which can be defined as crises, may arise along with the physical effects of the disease and the treatment process. It is suggested that the loss of dignity that develops in terminally ill patients causes the patients to want to die as soon as possible. It is important that patients receive care in accordance with the standards and value judgments they are used to, so that their sense of dignity and status is not affected by health problems. Dignity therapy is a type of short-term therapy developed to alleviate the distress of terminally ill patients and improve their end-of-life experiences. Chochinov emphasizes that dignity depends on productivity experiences, the search for purpose and meaning, defined dignity-protective care for patients facing a serious illness, and developed a model to be developed, studied and used by clinicians.

In the literature, it is seen that dignity therapy can be applied by different health professionals in patient groups with different diagnoses and provides positive contributions for patients and their relatives. With the increase in palliative care units in recent years, it has been considered important to apply this type of therapy to patients. In addition, no studies on dignity therapy have been found in Turkey. The aim of this study is to determine the effect of dignity therapy on the quality of life and depression levels of cancer patients.

Methods: The research was planned as a randomized controlled experimental study. Research Outpatient and inpatient treatment at Necmettin Erbakan University Faculty of Medicine hospital oncology clinic It will be done with end-stage cancer patients. October 2023-December 2023 with an average of 48 patients It will be carried out between . In collecting research data, Personal Information Form, Patient The Reputation Inventory and the Rosenberg Self-Esteem Scale (RSES) will be used.

Type of Research: Research, experimental, control group and pretest-posttest study will be carried out.

Place and Characteristics of the Research: The research was conducted in Konya province by Necmettin Erbakan It will be carried out in the Oncology clinic of University Meram Faculty of Medicine Hospital.Inpatient clinics are located on the 3rd and 4th floors, and there are 33 beds on each floor. Population of the Study: The population of the study was sent to Meram Medical Faculty Hospital Oncology Clinic consists of male and female inpatients.

Sample of the Research: Those who agreed to participate in the research and met the inclusion criteria. Patients who meet will be included in the study. The sample size in this study In order to determine the results, a priori power analysis was performed with the G-Power 3.1 statistical program. In determining the sample size, "The effect of Chinese culture-adapted dignity therapy on advanced cancer patients receiving chemotherapy in the Scores obtained from the "day oncology unit: A quasi-experimental study" study were used. 95% confidence (1-α), 80% test power (1-β), With an effect size of f = 0.78, the minimum number of samples to be included in the study was determined as 44 in total, 22 in each group. Patients are excluded from the study for many reasons. It was thought that there might be a loss of approximately 10% due to separation, and the number of samples was 48. It was planned to be.

Randomization: In this study, parallel group block randomization method was applied to the intervention and control groups. will be allocated randomly. Block randomization was used because the sample size was small. Patients will be selected equally using permutation method, and randomization will be selected using blocking technique. will be done. During randomization, CONSORT 2017 (Randomized Parallel Group Updated Guidelines for Reporting Research) will be used.

For randomization; To control for performance bias, patients will be blinded to the study hypothesis and will not be informed which group they are in. There will be no blinding for the researcher. However, blind technique will be used in the research. This blind technique will be applied by the researcher with the patients blinded until the application begins. In the research, in order to meet the blind technical conditions, the process steps were carried out by an independent statistician from the first stage. The sample will be sorted by a combination order and number. In this way selection bias will be controlled. The study will also be controlled for attrition bias and Statistics and reporting bias.

Data Collection Techniques and Tools: "Personal Information Form (sociodemographic and disease characteristics)", "Patient Dignity Inventory" and "Rosenberg Self-Esteem Scale" were used in data collection (RSES)" will be used.

Data Collection Tools Personal Information Form: The form created by the researcher by scanning the literature consists of 8 questions (age, gender, marital status, employment status, monthly income level, education level, cancer type, how long ago it was diagnosed).

Patient Dignity Inventory: The scale, consisting of a total of 25 items, was developed by Chochinov et al. (2008) and translated into Turkish by Eskigülek and Kav (2022) adapted. This five-point Likert type inventory is rated as "1 = no problem, 2 = slight problem, 3 = problem, 4 = big problem, 5 = very much problem." The minimum and maximum total score of the inventory is 25 and 125 points respectively. There are no reverse scored items in the inventory. A higher total score means that the individual's perceived reputation is complex. Items scoring three or more are clinically meaningful. As a result of factor analysis, a five-factor structure was obtained; The factors are reported as "symptom distress", "existential distress", "addiction", "peace of mind" and "social support". The Cronbach alpha value of the scale was reported as 0.94.

Rosenberg Self-Esteem Scale (RSES): The Rosenberg Self-Esteem Scale was developed by Morris Rosenberg in 1965 to measure the self-esteem of adolescents (Rosenberg, 1965). Participants score the questions as very true, true, false and very false. This scale, developed by Rosenberg, consists of a total of 63 items and 12 subtests. Self-Esteem Scale, one of these 12 subtests, was used in this study. The scale consists of a total of 10 items, 5 negative and 5 positive items. For questions 1, 2, 4, 6 and 7, respectively, it is very true (4), true (3), wrong (2), very wrong (1). The opposite is true for articles 3, 5, 8, 9 and 10. A high score on Rosenberg self-esteem means low self-esteem. A scale adaptation study was conducted by Çuhadaroğlu in 1985. As a result of this study, the test-retest reliability of the scale was found to be 0.75. The validity coefficient of the scale was found to be 0.71.

Application Steps: After the patients coming to the oncology clinic as outpatients or inpatients are evaluated by their physicians, they will be referred to the researcher if the predicted survival time is less than 6 months. The purpose of the study will be explained to patients who meet the inclusion criteria, and for those who accept, planning will be made in a way that will not disrupt the patient's treatment process, and the steps applied in dignity therapy will be followed. Dignity therapy will be applied in the interview room that will be requested in the oncology clinic to protect the confidentiality of information.

The application is planned as five sessions and the sessions will last approximately 40 minutes. Two questions in the dignity therapy protocol will be discussed in each session. Dignity Therapy Necmettin Erbakan University Faculty of Nursing, Department of Mental Health and Diseases Nursing. Lecturer It will be carried out by the researcher who serves as a member. She has worked as a clinical nurse researcher and is an expert in psychiatric nursing. Before the researcher started to apply this therapy, the 3-day "Dignity in Care - Online Training 2023" (https://www.cpd-umanitoba.com/events/dignityin-care-online-training) was held online between 14-28 September 2023. -2023/) attended the course. The course is hosted by Harvey Max Chochinov, a Distinguished Professor of Psychiatry at the University of Manitoba and Senior Scientist at the Cancer Care Manitoba Research Institute.

The therapist will interview each participant individually, it will be conducted in accordance with the dignity therapy protocol, the interviews will be recorded with a voice recorder, all recorded conversations will be transcribed and read to the patient after a preliminary arrangement.

A discussion will be held on the areas that the patient wishes to change in the text, and as included in the dignity therapy protocol, a session organization process will be carried out with the participant, especially in the last session, in which the participant will be provided with a written legacy (certificate of productivity). The Dignity therapist prepares a document to be transferred to the participants' families, relatives or friends, with patient approval. It will be made ready to be given after submission. The Dignity therapist will create a written report at the end of the interviews to be given to their families and present this report to the patients. The final version of the report will be given by the patients.

Data Collection: Data will be collected by the researcher through face-to-face interviews in the oncology clinic at Necmettin Erbakan University Faculty of Medicine Hospital, from patients who meet the inclusion criteria and agree to participate in the study, without disrupting the working order of the clinic. Data collection forms will be applied to both the experimental and control groups as a pretest before dignity therapy begins to be applied to the participants (in the 1st session) and as a posttest after dignity therapy is completed (in the last session). Data collection tools will be filled in the patient room, respecting the patient's privacy.

Research Variables Dependent variables: Patient Dignity Inventory, Rosenberg Self-Esteem Scale Independent variables: Sociodemographic and disease characteristics, applied dignity therapy Control variables: Age, gender Ethical Dimension of the Research: Permission for the research was received from Necmettin Erbakan University Health Sciences Scientific Research Ethics Committee and the Faculty of Medicine Hospital Oncology Clinic. Permission will be obtained via e-mail from the authors of the scales to be used. Participants who will participate in the research will be given verbal information about the research and Informed Consent Form will be signed.

Participants who do not agree to participate in the research will not be forced to participate. There is no conflict of interest between the researchers.

Statistical Evaluation of Data: Statistical analysis will be done using SPSS 23.0 (Statistical Package for Social Sciences Version 23.0) program. Cronbach's Alpha analysis will be used in the internal consistency examination to determine the validity and reliability of the scale, descriptive statistics will be used to determine the findings regarding the individual characteristics of the participants, median and minimum/maximum values for non-normally distributed variables, and mean±standard deviation values for normally distributed variables. Appropriate statistical analyzes regarding the hypotheses will be used to compare independent variables. The results obtained will be tested at the p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Participants in the Study:

  * Able to speak and understand Turkish,
  * Those over 18 years of age
  * No communication barriers
  * Cancer diagnosis is in the 4th stage and in the last stage
  * Patients with a predicted survival time of less than 6 months (physician opinion) will be included

Exclusion Criteria:

* Criteria for Exclusion of Participants in the Study:

  * Those diagnosed with dementia, delirium or other organic brain disorders;
  * Those with impaired consciousness;
  * Patients with mental problems that prevent them from receiving esteem therapy will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient Dignity Inventory | first week and within one week after completion of therapy
  The scale, consisting of a total of 25 items, was developed by Chochinov et al. (2008) and translated into Turkish by Eskigülek and Kav (2022) adapted. The minimum and maximum total score of the inventory is 25 and 125 points respectively. There are no reverse scored items in the inventory. A higher total score means that the individual's perceived reputation is complex. Items scoring three or more are clinically significant. As a result of factor analysis, a five-factor structure was obtained; The factors are reported as "symptom distress", "existential distress", "addiction", "peace of mind" and "social support"

SECONDARY OUTCOMES:
Personal Information Form | first week and within one week after completion of therapy
  The form created by the researcher by scanning the literature consists of 8 questions
Rosenberg Self-Esteem Scale | within one week after completion of therapy
  The Rosenberg Self-Esteem Scale was developed by Morris Rosenberg in 1965 to measure the self-esteem of adolescents (Rosenberg, 1965). Participants score the questions as very true, true, false and very false. This scale, developed by Rosenberg, consists of a total of 63 items and 12 subtests. Self-Esteem Scale, one of these 12 subtests, was used in this study. The scale consists of a total of 10 items, 5 negative and 5 positive items. A high score on Rosenberg self-esteem means low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: NESIBE GÜNAY MOLU, Principal Investigator — Necmettin Erbakan University

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to protection of patient confidentiality and institutional rules.